CLINICAL TRIAL: NCT04798248
Title: Evaluation of Momentary Affect Regulation - Safer Sex Intervention
Acronym: MARSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 TP2AH000076-01-00
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Momentary Affect Regulation - Safer Sex Intervention (Experimental): Momentary Affect Regulation - Safer Sex Intervention (MARSSI) is the treatment condition. MARSSI aims to enhance an individual's motivation to change risk behaviors, provides skills to address depression's effects on behavior, and prompts and reinforces healthy affect regulation, cognitive behavioral skill use, and behavior change in daily life.
  Interventions: Behavioral: Momentary Affect Regulation - Safer Sex Intervention (MARSSI)
- Podcast Health Group (Sham Comparator): The Podcast Health Group is the control counterfactual condition.
  Interventions: Behavioral: Podcast Health Group

INTERVENTIONS:
Behavioral: Momentary Affect Regulation - Safer Sex Intervention (MARSSI) — MARSSI is an individual-level intervention that involves a one-hour manualized session with a sexual reproductive health (SRH) counselor, followed by one-month of daily use of a mobile health app and a final 20-minute booster session with the SRH counselor.
  Arms: Momentary Affect Regulation - Safer Sex Intervention
Behavioral: Podcast Health Group — Participants assigned to the Podcast Health Group will listen to ~20 minute podcast episode put out by the Susan G. Komen Foundation about family history of breast cancer; the podcast does not include information related to the outcomes of interest for the study.
  Arms: Podcast Health Group

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in the Momentary Affect Regulation - Safer Sex Intervention (treatment) relative to the offer to participate in the control condition on participants' reported condom use, use of effective contraception, and number of sexual partners three months after the end of the treatment intervention.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be conducting a rigorous evaluation of an innovative intervention designed to reduce unplanned pregnancy and sexually transmitted infections in young women with depression, entitled Momentary Affect Regulation - Safer Sex Intervention (MARSSI). MARSSI was developed by Dr. Lydia Shrier of Boston Children's Hospital. MARSSI has three components. The first is a manualized session with a sexual and reproductive health counselor, who uses motivational interviewing (MI) techniques to help the young woman identify a risk-reducing goal for her sexual behavior, develop a change plan, and provide depression education and skills, based on cognitive behavioral therapy. The second component is a mobile health (mhealth) application that the young woman loads on her smartphone and, for four weeks, uses to complete app-prompted reports 3 times a day and a scheduled report once a day. When she reports poor affect, low contraceptive or condom self-efficacy, pregnancy desire, or desire for sex to regulate affect, she receives personalized messages prompting healthy behaviors and cognitive behavioral skill use. The third component is a booster session that occurs after 4 weeks of app use. The young woman meets with the counselor again to review her behavior and relationships, discuss progress toward her goal, and learn a new skill. Through these components, MARSSI aims to enhance motivation to change risk behaviors, provides skills to address depression's effects on behavior, and prompts and reinforces healthy affect regulation, cognitive behavioral skill use, and behavior change in daily life.

The Policy & Research Group (PRG) will conduct an implementation evaluation and an impact evaluation, using an individual randomized controlled trial, to test the efficacy of this new intervention. The study will target young women ages 16-21 who have depressive symptoms and are recent clients of sexual and reproductive health clinics. The primary focus of the study will be to investigate the impact of the intervention on three self-reported sexual behaviors: 1) condom use; 2) use of effective contraception; and 3) number of sexual partners. The study will also include exploratory investigations of a number of other sexual behaviors and theoretically relevant antecedents to change in behavior and sexual health, including but not limited to: 1) engagement in protective sexual behavior; 2) condom use at last vaginal sex; 3) effective contraceptive use at last vaginal sex; 4) dual methods of protection; 5) frequency of vaginal, anal, and oral sex; 6) substance use before any type of sex; 7) types of sexual partners/relationships; 8) depressive symptoms; 9) sexual communication self-efficacy; 10) motivation to change risky sexual behaviors; 11) contraceptive and condom knowledge; 12) contraceptive and condom planning self-efficacy; and 13) use of cognitive restructuring.

Outcomes will be assessed using self-reported, participant-level data gathered (by way of a questionnaire) at four time points: baseline (enrollment); post-program (immediately after the end of the intervention period; 1 month post baseline); short-term (4 months post-baseline) follow-up; and long-term (7 months post baseline) follow-up.

Starting in June 2021 and continuing for 23 months, 600 participants who have received reproductive health care in the past two years (nationally) will be recruited and enrolled into the study by trained Planned Parenthood research coordinators. The final year of the grant will be used to complete the following tasks: collect follow-up data from study participants; conduct implementation and impact evaluation analysis, reporting, and dissemination efforts; and manualize and package the curriculum and training materials.

ELIGIBILITY:
Inclusion Criteria:

* Visited reproductive health care provider in the past two years
* Own a smartphone
* Have the technical capacity to participate
* Be fluent in English
* Be 16 to 21 years of age
* Be biologically able to become pregnant (to the best of their knowledge)
* Score at least 8 on the PHQ-8
* Have had penile-vaginal sex in the past 3 months
* Have had penile-vaginal sex at least once a week, on average
* Report having done at least one of the following during the 3 months preceding eligibility screening: 1) Not using a condom every time they have sexual intercourse; 2) Used condoms, a diaphragm, cervical cap, spermicide, sponge, fertility awareness, or withdrawal as a primary form of birth control; 3) Had sexual intercourse with more than one person; 4) Had sexual intercourse within 2 hours after using drugs and alcohol; and/or 5) Been treated for an STI/STD

Exclusion Criteria:

* Trying to get pregnant or currently pregnant at the time of eligibility screening
* Have given birth during the 6 months preceding eligibility screening
* Married or engaged to be married at the time of eligibility screening
* Identified as fraudulent

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Be biologically able to become pregnant (to the best of their knowledge)
Enrollment: 405 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Times having vaginal sex without a condom | Assessed three months after the intervention period has ended
  Participant self-report on the number of times having vaginal sex without using a condom during the past 30 days
Number of sexual partners | Assessed three months after the intervention period has ended
  Participant self-report of the number of sexual partners in the the past three months
Effective contraceptive use | Assessed three months after the intervention period has ended
  Participant self-report on whether or not they are currently using effective (prescription) contraception or not

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, Principal Investigator — The Policy & Research Group
Locations (2):
- United States (2):
  - Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky, Seattle, Washington
  - Planned Parenthood of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.
Access Criteria: For any individuals interested in accessing a copy of this public use dataset, please email info@policyandresearch.com with your inquiry.
URL: https://acrobat.adobe.com/id/urn:aaid:sc:VA6C2:848c078d-7652-4647-b19c-94f97efb1f2e

REFERENCES:
- Available data/document: Information on publicly available dataset — https://acrobat.adobe.com/id/urn:aaid:sc:VA6C2:e0548c67-55a8-452d-9854-ade3876c29d8 — For any individuals interested in accessing a copy of this public use dataset, please email info@policyandresearch.com with your inquiry.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT04798248/SAP_001.pdf